CLINICAL TRIAL: NCT03906032
Title: Prospective Randomized Controlled Comparison of Sliding Hip Screw to Intra Medullary Nailing in the Treatment of Intertrochanteric Hip Fracture
Brief Title: Comparison of Sliding Hip Screw to Intra Medullary Nailing in the Treatment of Intertrochanteric Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Waterford (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, May Cleary, PI, University Hospital Waterford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHWHip#
Record Dates: First submitted 2019-04-01; First posted 2019-04-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hip Fractures; Gait, Unsteady; Function
Keywords: Timed up and go; mobility; functional outcome
MeSH Terms: conditions — Hip Fractures; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Gait speed (mean velocity): Sample size calculations are based on a two-sample, two-sided t-test for a difference in means with 80% power, a 5% type 1 error rate. The minimal clinically important difference (MCID) in gait speed is stated in the literature as between 0.10 - 0.20 m/s. We considered treatment effect of 0.2 m/s (while assuming a SD of 0.3). The resulting total sample sizes for this effect is 74 patients at the 6 months post-operative timeframe. A significant attrition rate (50%) for this population will be allowed for by additional recruitment of >150 participants
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Simple randomization technique using an online random number generator will be utilized. Sequential sealed envelopes with group allocation will be opened at the time of the daily trauma meeting and the appropriate plan made for the patient. Patients are randomized according to 3 mobility groups - independent, walking stick/crutch or walking frame.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-medullary hip Nail (Experimental): Surgery
  Interventions: Device: TFNA IM Nail
- Sliding hip screw (Active Comparator): Surgery
  Interventions: Device: Sliding hip screw

INTERVENTIONS:
Device: TFNA IM Nail — IM nail
  Arms: Intra-medullary hip Nail
Device: Sliding hip screw — SHS surgical fixation
  Arms: Sliding hip screw

SUMMARY:
Shortening of the abductor lever arm is a particular concern with the SHS, and the resultant biomechanical alterations may impair gait, including decreased cadence, gait speed and increased double support time on the injured side.

The use of an IM nail device may reduce shortening and improve functional parameters in this patient cohort

DETAILED DESCRIPTION:
Published work in this field to date has not demonstrated an advantage of nailing over hip screw in intertrochanteric proximal femoral fractures. The current literature focus on outcome questionnaires, pain scores and basic functional tests alone may not delineate all functional benefits. A key factor in whether a person, post hip fracture, returns to independent living is gait speed. The cost implications on the healthcare provider of having 30% of this ever increasing group losing their independence and requiring admission to a care facility post hip fracture is a growing problem.

Shortening of the abductor lever arm is a particular concern with the SHS, and the resultant biomechanical alterations may impair gait, including decreased cadence and increased double support time on the injured side.

The cost differential between a nail and a SHS is a barrier to routine use of nailing in this population unless a clear benefit is demonstrated. Fracture nonunion is uncommon in this injury however improving functional outcome and reducing morbidity and mortality in this group is important.

In this prospective randomised study, the investigators examine whether an intramedullary nail (TFNA) results in a greater functional benefit in A1/A2 intertrochanteric fractures compared with the SHS, in terms of gait speed and other objective gait assessments, as well as other established post operative outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* OTA Hip fracture grade A1 and A2
* Greater than 18 years old

Exclusion Criteria:

* Fracture less than 18 yrs old
* Fracture with lateral wall trochanteric comminution
* Poltrauma
* Concurrent lower limb fractures
* Immobile/wheelchair/bedbound patients
* High energy hip fractures
* Pathological fractures
* Reverse oblique and sub-trochanteric femoral fractures which are considered obligate TFNA at our centre
* Open wounds on affected limb
* Active psoriasis or other dermatological conditions at affected area
* Unable to gain consent from patient or patient's NOK

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Kinmeatic Gait parameters at Hip | 6 months
  Rate of change in hip kinematic profile between baseline and subsequent time points,

SECONDARY OUTCOMES:
Length of stay | Through to study completion at one year post operatively.
  The duration of hospital stay after this procedure has wide variability between 3 days and weeks to months.
Change in Heamoglobin concentration post surgery | Day 2 post surgery
  Haemoglobin (Hb) day two measurement in grams per decilitre (g/dl)
Change in Heamatocrit concentration post surgery | Day 2 post surgery
  Haematocrit day two measurement in litre of cells per litre of blood (L/L)
Mortality | At any time point to 1 year post op
  Absolute
Analgesia Use | 5 days
  rate of opiate use
Timed up and go test | 6 weeks, 6 months, 1 year
  Tested measure of mobility and the change between baseline and subsequent time points
Harris Hip score | 6 weeks, 6 months, 1 year
  Functional scale of hip pain and the change between baseline and subsequents time points. Maximum score: 100 points indicating excellent function, minimum score 0 points indicating poor function
Radiographic assessment of fracture healing | 6 weeks, 6 months, 1 year
  Radiographic union as observed on plain radiographs at the stated time intervals (radiographic union score for hip total score of 10 - 30 points, minimum 10, maximum 30)
Radiographic assessment of femoral neck shortening | 6 months
  Radiographic assessment of any change in femoral neck length (in millimetres) between image on date of surgery and the 6 month post surgery image

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Waterford, Waterford, Ireland

IPD SHARING:
Plan to Share IPD: No